CLINICAL TRIAL: NCT06414655
Title: Multicenter Prospective Cohort Study of Twin Maternal-Child Dyads in China
Acronym: ChiTwiMC
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Chongqing Medical University (Other); Shengjing Hospital (Other); Peking University (Other); Nankai University (Other); Shanghai First Maternity and Infant Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); International Peace Maternity and Child Health Hospital (Other); The Second Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ChiTwiMC
Record Dates: First submitted 2024-03-17; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-01

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication; Twin to Twin Transfusion as Antepartum Condition; Pre-Term; Pre-Eclampsia; Twin Monochorionic Diamniotic Placenta; Twin Dichorionic Diamniotic Placenta; High Risk Pregnancy; Twin Placenta
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Collecting peripheral venous blood from husband, hair during the first trimester, peripheral venous blood and cervicovaginal secretions during the first trimester, second trimester, late pregnancy before labor, placental tissue, amionic fluid and umbilical cord blood during delivery, hair, meconium of newborns, and buccal mucosa from infants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter Prospective Cohort Study of Twin Maternal-Child Dyads in China (ChiTwiMC) is supported by National Key Research and Development Program of China - Reproductive Health and Women's and Children's Health Protection Project. This project is funded by the Ministry of Science and Technology of China under grant number 2023YFC2705900. The ChiTwiMC cohort is led by Professor Wei Yuan from the Department of Gynecology and Obstetrics at Peking University Third Hospital.

DETAILED DESCRIPTION:
The ChiTwiMC Cohort focusing on the serious complications of twin pregnancy, establish a multicenter large prospective mother-child cohort of twin pregnancy covering pregnancy→neonatal period→early childhood, and a multi-variety, multi-stage biobank for the study of adverse outcomes of twin pregnancy. The ChiTwiMC Cohort is planning to recruit 2000 pregnant women aged 18-45 years from 9 large obstetrical center of major University-affiliated Hospitals across China, between December 2023 and May 2026. All women will be enrolled prior to 14 wks of gestation, pregnancy was followed up at 22-28 wks, 30-38 wks of gestation, delivery, postpartum 42 days, 6 months, 12 months. Data including demographics, medical history, reproductive history, clinical diagnosis, treatment information, and pregnancy and birth outcomes will be collected via electronic data capture system. Track the outcome of severe maternal-fetal complications and early neonatal outcomes of twins, and collect biological samples, including peripheral venous blood, hair and cervicovaginal secretions from pregnant women, placenta tissue, amniotic fluid and unbilical cord blood at delivery, meconium and hair from newborns, buccal mucosa from infants and peripheral venous blood from the husband.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancies
* Female aged between 18-45 years
* Gestational age is less than 14 weeks
* Planning to receive prenatal healthcare and delivery service at the study hospital
* Signing informed concent and willing to participate

Exclusion Criteria:

* Women with mental disorders or serious maternal illness that is not eligible to participate
* Inability to provide informed consent
* Pregnant women not registered in our hospital

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The ChiTwiMC is a prospective cohort that will enroll 2000 pregnant women aged 18-45 years and over from 9 large obstetrical centers of University-Affiliated Hospitals (Peking University Third Hospital; First Affiliated Hospital, Sun Yat-Sen University; Chongqing Medical University; Shengjing Hospital; Shanghai First Maternity and Infant Hospital; The First Affiliated Hospital of Anhui Medical University; International Peace Maternity and Child Health Hospital; The Second Hospital of Shandong University; Shandong Provincial Hospital). These hospitals located at 7 supercities (Beijing, Shanghai, Guangzhou, Shenyang, Jinan, Chongqing, and Hefei) of China. Pregnant women who are planning to receive prenatal healthcare and delivery in those hospitals are potential candidates for the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of preterm delivery | From inclusion to delivery
  Preterm delivery is defined as delivery between 28 and 37 gestational weeks.
Rate of preeclampsia | From inclusion to delivery
  Preeclampsia is defined as the condition occurring in pregnant women after 20 weeks of gestation, characterized by systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, accompanied by any of the following: a urinary protein quantification ≥0.3 g/24 h, or a urine protein/creatinine ratio ≥0.3, or random urine protein ≥ (+) (as a method of examination when protein quantification is not feasible). In the absence of proteinuria, the condition may still be diagnosed if there is involvement of any organ or system, including but not limited to critical organs such as the heart, lungs, liver, kidneys, or abnormalities in the hematological, digestive, or neurological systems, as well as complications affecting the placenta-fetus.
Rate of twin-to-twin transfusion syndrome (TTTS) | From inclusion to delivery
  TTTS is diagnosed in monochorionic diamniotic twin pregnancies when there is a discordance in amniotic fluid volumes, with one fetus exhibiting polyhydramnios and the other oligohydramnios. Specifically, before 20 weeks of gestation, the condition is diagnosed if one fetus (the recipient) has a deepest vertical pocket (DVP) of amniotic fluid ≥8cm, while the other fetus (the donor) has a DVP ≤2cm; after 20 weeks of gestation, the diagnosis is made if one fetus (the recipient) has a DVP ≥10cm, while the other fetus (the donor) has a DVP ≤2cm.
Rate of selective fetal growth restriction (sFGR) | From inclusion to delivery
  sFGR is diagnosed in monochorionic diamniotic twin pregnancies when one fetus has an estimated fetal weight below the 10th percentile for its gestational age, and there is a discrepancy of ≥25% in the estimated fetal weights between the two fetuses.
Rate of fetal brain injury | From inclusion to delivery
  Fetal brain injury is an abnormality in the structural and functional integrity of the cerebrum, cerebellum, or brainstem during the gestational period, caused by various factors such as hypoxic-ischemic events, infections, hemorrhage, congenital malformations, and genetic metabolic disorders.
Rate of neonatal brain injury | From inclusion to delivery
  Brain injury refers to damage to the central nervous system resulting from various risk factors during pregnancy, childbirth, and the neonatal period. Clinically, it manifests as central motor disorders, cognitive impairments, language disorders, visual and auditory impairments, as well as difficulties in social interaction and psychological and behavioral disorders. It needs pregnant history or birth history, (such as one of twin intrauterine fetal death, Intrauterine distress), manifestation, and ultrasound, CT, MRI, electroencephalogram to make a definite diagnosis.
Rate of early childhood developmental delay of the offspring | Within 1 year after delivery
  Early childhood developmental delay of the offspring refers to a significant lag or delay in achieving age-appropriate developmental milestones across one or more domains, including cognitive, language, motor, social-emotional, and adaptive skills, during the early years of life (typically from birth to 5 years of age) in comparison to established norms or peers. The assessment of early childhood developmental delay is conducted using standardized scales such as Ages Stages Questionnaires (Third Edition), Gesell Developmental Schedules, and Bayley Scales of Infant and Toddler Development. The actual measurement process will be depending on the routine pediatric settings and resources available at each participating institution.
Children's height | Within 1 year after delivery
  Each child is measured twice. If the difference is less than 0.1 cm, the average of the two measurements is taken. If the difference is greater than 0.1 cm, the measurement is repeated.
Children's weight | Within 1 year after delivery
  Each newborn is measured twice. If the difference is less than 0.01 kg, the average of the two measurements is taken. If the difference is greater than 0.01 kg, the measurement is repeated.

SECONDARY OUTCOMES:
Rate of sleep disorders | From inclusion to delivery
  Women's physiological and psychological changes during pregnancy will affect sleep, and the occurrence of bad sleep during pregnancy is more common. It is generally assessed by a sleep questionnaire.
Rate of mental and phycological disorders | From inclusion to delivery
  Maternal mental health is as important as physical health, and good maternal mental health helps to promote the physical and mental health of the baby, as well as their own physical condition and natural childbirth. The condition of pregnant women is generally assessed by psychiatric departments.
Rate of single intrauterine fetal demise | From inclusion to delivery
  The death of one fetus for twin pregnancy，the occurrence in the second and third trimesters of pregnancy has substantial adverse effects on surviving infants.
Rate of gestational hypertension | From inclusion to delivery
  Take two consecutive measurements on the same arm, the systolic blood pressure more than 140 mmHg and (or) the diastolic blood pressure more than 90 mmHg. High blood pressure may lead to severe complications such as preclampsia and clampsia.
Rate of gestational diabetes mellitus | From inclusion to delivery
  Diagnosed with gestational diabetes through an oral glucose tolerance test (OGTT). The blood glucose threshold of fasting, 1 h and 2 h after taking oral glucose was 5.1, 10.0, 8.5 mmolL, respectively, and the blood glucose level reached or exceeded the above criteria at any time point was diagnosed as GDM. GDM is clearly associated with adverse pregnancy outcomes such as fetal macrosomia, cesarean section delivery, preterm birth, and preeclampsia
Number of maternal death | From inclusion to delivery
  Deaths during pregnancy or less than 42 days after termination of pregnancy.
Rate of stillbirth | From inclusion to delivery
  After 28 gestational weeks, the fetus dies before or during delivery
Birth weight | At delivery
  Each newborn is measured twice. If the difference is less than 0.01 kg, the average of the two measurements is taken. If the difference is greater than 0.01 kg, the measurement is repeated.
Birth length | At delivery
  Each newborn is measured twice. If the difference is less than 0.1 cm, the average of the two measurements is taken. If the difference is greater than 0.1 cm, the measurement is repeated.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Wei, PhD, MD, Study Chair — Obstetrics and Gynecology Department of Peking University Third Hospital
Locations (11):
- China (11):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University, Beijing, Beijing Municipality
  - Chongqing Medical University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shengjing Hospital, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - International Peace Maternity and Child Health Hospital, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - Nankai University, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
We have decided that the program will be confidential and not open to other researchers